CLINICAL TRIAL: NCT00660400
Title: A Pilot Study Of Pre-Transplant 5-Azacitidine (Vidaza) In Patients With High-Risk Myelodysplastic Syndrome (MDS) Who Are Candidates For Allogeneic Hematopoietic Cell Transplantation
Brief Title: Pre-Transplant 5-Azacitidine In Patients With High-Risk Myelodysplastic Syndrome Who Are Candidates For Allogeneic Hematopoietic Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15158; 106349 (Other: USF IRB)
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia
Keywords: Myeloid; Monocytic
MeSH Terms: conditions — Leukemia | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Therapy (Experimental): 5-azacitidine therapy followed Allogeneic Hematopoietic Cell Transplantation (HCT).
  Interventions: Drug: 5-azacitidine; Procedure: Allogeneic Hematopoietic Cell Transplantation (HCT)

INTERVENTIONS:
Drug: 5-azacitidine — Once enrolled, the patients will receive pre-transplant 5-azacitidine (Vidaza) 75 mg/M^2/day subcutaneously for 5-7 days every 28 days). Adjustments in dose and timing may occur based on clinical and hematological parameters.
  Other Names: Vidaza
Procedure: Allogeneic Hematopoietic Cell Transplantation (HCT) — Patients will receive transplantation if there is either a suitable sibling or an unrelated donor.
  * Response will be evaluated by bone marrow biopsy after 4 cycles of 5-azacitidine or prior to HCT whichever comes first. Due to the very high risk of progression to AML or death in this patient population, the HCT will be done as soon as possible.
  * The patients may have additional cycles of 5-azacitidine per standard hematology practice until scheduled for transplant or until progression of disease.
  * All patients will be followed until time to progression of MDS, AML or death or a maximum of 1 year. For patients that are transplanted, follow up will be to one year post-transplant.
  Other Names: HCT

SUMMARY:
The purpose of this study is to find out if treating people who have high-risk myelodysplastic syndrome (MDS) with 5-Azacitidine (Vidaza) prior to their allogeneic hematopoietic cell transplant (HCT) is helpful in preventing their myelodysplastic syndrome from coming back.

In previous research, 5-Azacitidine appeared to help the bone marrow of a patient with MDS begin to function more normally. This means bone marrow cells can grow and do their work the way they were meant to. 5-Azacitidine is approved by the Food and Drug Administration (FDA) for the treatment of MDS. The effect of 5-Azacitidine in patients receiving hematopoietic cell transplants have not been studied.

DETAILED DESCRIPTION:
RESEARCH PLAN

* This will be a single-center prospective trial
* Patients with high risk MDS that are potentially eligible for HCT will be enrolled.
* A donor search will be initiated, and 5-Azacitidine will be given per standard practice.
* 5-Azacitidine dose is 75 mg/M^2/day subcutaneously by standard practice (generally this is 7 days per monthly cycle, but alterations occur depending on clinical and laboratory parameters).
* Patients where a suitable donor is not found can continue with 5-Azacitidine per standard treatment. These patients will be followed until progression of MDS to acute myelogenous leukemia (AML) or death, for up to one year.
* If a suitable donor is obtained, the patient will proceed to HCT. The HCT conditioning regimen will be dictated by the Blood and Marrow Transplant (BMT) physician. While waiting HCT, additional cycles 5-Azacitidine may be given. Pre-HCT conditioning regimen therapy will begin no more than 8 weeks and no less than 4 weeks after the last administration of 5-Azacitidine.
* As the number of cycles of 5-Azacitidine is not standardized and the retrospective review of our patients noted above indicated a benefit to ANY exposure to 5-Azacitidine, the actual number of cycles of 5-Azacitidine delivered will not be specified. In addition, as high risk MDS patients have an average time to death of 0.4 years, any delay to HCT once it is available is to be avoided.
* A bone marrow biopsy will be performed to reassess disease response to therapy after the last cycle of 5-Azacitidine before transplant, or after the fourth cycle of 5-Azacitidine, whichever comes first. Note that both the biopsy and the timing of the biopsy is a standard evaluation procedure.
* Donor progenitor cell collection will be prescribed by the BMT Attending Physician.

HCT

* The patient will undergo HCT designated per attending BMT physician.
* Supportive care will be based on institutional guidelines, Stem cell collections, processing and laboratory studies

Stem cell collections, processing and laboratory studies

* Graft assessment, processing, and characterization will be done as per institutional guidelines
* Chimerism testing will be obtained to document post-transplant engraftment, per standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Potential candidate for HCT.
* Histologically confirmed diagnosis by pathologic review of previous diagnosis of high-risk myelodysplastic syndrome (MDS): International Prognostic Scoring System (IPSS) > 1 or AML-MDS or treatment related MDS.
* Serum bilirubin levels ≤1.5 times the upper limit of the normal (ULN) range for the laboratory. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis; Serum glutamic-oxaloacetic transaminase (SGOT) [aspartate aminotransferase (AST)] or serum glutamic pyruvic transaminase (SGPT) [alanine aminotransferase (ALT)] levels ≤2 x ULN.
* Serum creatinine levels ≤1.5 x ULN
* Karnofsky performance status greater or equal to 70%
* Signed informed consent form in accordance with institutional policies

Exclusion Criteria:

* Known or suspected hypersensitivity to Vidaza or mannitol
* Pregnant or lactating women
* Human immunodeficiency virus (HIV) or seropositive, confirmed by nucleic acid amplification testing (NAT)
* Active central nervous system (CNS) malignancy
* Active infection
* History or presence of primary hepatoma

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Field, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Janelle Perkins, Pharm.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Nishihori T, Perkins J, Mishra A, Komrokji R, Kim J, Kharfan-Dabaja MA, Perez L, Lancet J, Fernandez H, List A, Anasetti C, Field T. Pretransplantation 5-azacitidine in high-risk myelodysplastic syndrome. Biol Blood Marrow Transplant. 2014 Jun;20(6):776-80. doi: 10.1016/j.bbmt.2014.02.008. Epub 2014 Feb 15. PMID 24534108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 05/2008 to 08/2010, 25 patients with Myelodysplastic Syndrome (MDS) were enrolled to the study at Moffitt Cancer Center.
Pre-assignment Details: Four patients did not proceed to allogeneic HCT.
Period: Overall Study
Arm/Group | Combined Therapy
Started | 25
Completed | 21
Not Completed | 4
Not completed — Lack of insurance approval | 1
Not completed — Suboptimal organ function | 1
Not completed — Intracranial hemorrhage | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 21 of 25 participants proceeded to allogeneic HCT and were evaluated for most measures.
Arm/Group | Combined Therapy
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 67]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse-free Survival (RFS)
Description: Relapse-free survival one year after allogeneic HCT in MDS patients receiving at least one complete cycle of 5-azacitidine (Vidaza) in the pre-transplantation setting. Relapsed disease: if with complete remission (CR) - greater than 5% blasts in bone marrow; if with partial response (PR) - greater than 30% increase in blasts in the marrow; if with stable disease (SD) - return to pretreatment peripheral blood levels and transfusion requirements due to disease.
Time Frame: One year post allogeneic HCT
Population: Participants who proceeded to allogeneic HCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Therapy
Number analyzed (Participants) | 21
percentage of participants | 52 [30 to 71]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Pre-allogeneic HCT responses to 5-azacitidine (Vidaza), based on the International Working Group criteria: Complete Remission (CR); Partial Response (PR); Stable Disease (SD). Point estimates and 95% confidence intervals were calculated for the response rate to 5-azacitidine, evaluated at marrow evaluation after 4 cycles of 5-azacitidine or prior to HCT whichever came first. CR: Bone marrow with 5% myeloblasts and normal maturation of all cell lines. PR: All CR criteria if abnormal before treatment except bone marrow blasts decreased by 50% over pretreatment but still > 5%. SD: Failure to attain CR, PR, relapsed (or progressive) disease.
Time Frame: At the end of up to six (28 day) cycles of 5-azacitidine
Population: Participants who proceeded to allogeneic HCT
Measure: Number; unit: percentage of participants
Arm/Group | Combined Therapy
Number analyzed (Participants) | 21
percentage of participants
  Partial Response | 48
  Complete Remission | 0
  Stable Disease | 33
  Progressive Disease | 19

3. Secondary Outcome: Percentage of Participants Who Proceed to Hematopoietic Cell Transplantation (HCT)
Description: Proportion of patients enrolled who subsequently proceeded to allogeneic HCT.
Time Frame: Up to 3 years
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Combined Therapy
Number analyzed (Participants) | 25
percentage of participants | 84

4. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival for all participants at one year after first dose of 5-azacitidine (Vidaza). Overall survival was calculated by the method of Kaplan-Meier with standard errors computed using Greenwood's formula.
Time Frame: One year
Population: Participants who proceeded to allogeneic HCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Therapy
Number analyzed (Participants) | 21
percentage of participants | 62 [38 to 79]

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Description: This was a standard of care study for Myelodysplastic Syndrome patients, with 5-Azacitidine prior to standard transplant.
Arm/Group | Combined Therapy
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Therapy (N=25)
Constitutional symptoms - Other, fatigue (General disorders) | 1 (1)
Constitutional symptoms - Other, anorexia (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) - skin (cellulitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1)
Creatinine - Acute renal failure (Metabolism and nutrition disorders) | 1 (1)
Neurology - Other, weakness (Nervous system disorders) | 1 (1)
Neurology - Other - numbness, tingling (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other, pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Infection - Other, sepsis (Infections and infestations) | 1 (1)
Deep venous thrombosis (Vascular disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitation: Small single center pilot study to show the use of pre-treatment 5-Azacitidine and successfully proceeding to transplant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes